CLINICAL TRIAL: NCT06102798
Title: The Efficacy and Safety of Acupuncture in Relieving Neurogenic Claudication Among Patients With Lumbar Spinal Stenosis: a Randomized Controlled Trial
Brief Title: Acupuncture for Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-039-KY-01
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Acupuncture; Neurogenic Claudication; Randomized controlled trial; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Hwato brand disposable acupuncture needles and adhesive pads will be used. The acupoints of Shenshu (BL23), "Dachangshu (BL25)", Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be inserted. There will be 18 treatment sessions with 3 times a week for continuous 6 weeks and a 30 min treatment per session.
  Interventions: Device: Acunpuncture
- Sham acupuncture (Sham Comparator): Hwato brand disposable placebo needles (with the handle identical to the needles in the acupuncture group and the body at a size 0.30 × 25 mm) and adhesive pads will be used. The acupoints of Shenshu (BL23), Dachangshu (BL25), Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be selected. The treatment duration and frequency of sessions for participants in the SA group will be the same as in the acupuncture group.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acunpuncture — For the bilateral" BL25", sterile disposable steel needles (Hwato, China; 0.3 mm×75 mm) will be inserted through adhesive pads to a depth of 50-70mm until participates feel a sensation similar to electric shock radiating downward to the knees. For the other four acupoints (BL23, BL40, BL57 and KI3), the needles (Hwato, China; 0.3 mm×40 mm) will be inserted through adhesive pads to a depth of 15-25 mm, gently rotated three times and lifted to achieve de qi.
  Arms: Acupuncture
Device: Sham acupuncture — For all the points, the needles will be inserted into adhesive pads without skin penetration. Needles will be lifted, thrust and twirled for 3 times to mimic real acupuncture. No manipulation will be conducted during 30-minute maintenance.
  Arms: Sham acupuncture

SUMMARY:
The clinical trial aims to evaluate the efficacy and safety of acupuncture in alleviating neurogenic claudication symptoms among patients with degenerative lumbar spinal stenosis (LSS).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnosis criteria of LSS;
2. Aged between 50-80 years;
3. Neurogenic claudication (NC) for more than 3 months;
4. Able to walk for at least 20 meters continually without device assistance, and forced to stopped walking out of NC within 30 mins in the meanwhile;
5. The average pain of buttocks and/or legs scores≥4 on the Numerical Rating Scale (NRS) when walking, standing, or extending the back in the past week;
6. More severe pain in the buttock and/or leg than in the lower back;
7. Score at least 7 on Modified Roland-Morris Disability Questionnaire（RMDQ）;
8. Central sagittal diameter stenosis of lumbar spinal canal as manifested by MRI or CT scan;
9. Volunteer to participate the trial and provide written informed consent.

Exclusion Criteria:

1. Non-degenerative LSS, such as congenital, post-traumatic or spondylolisthesis LSS; operation indications, such as segmental muscular atrophy, bowel and bladder disfunction, and spinal instability; tuberculosis or tumor in the lumbar area; or multiple vertebral compression fracture or compression fracture in the segment of stenosis;
2. Vascular claudication;
3. Severe heart, pulmonary, liver and/or kidney diseases;
4. Clinical comorbidities that may interfere with the assessment of pain intensity or walking ability, such as fibromyalgia, chronic widespread pain, amputation, stroke, Parkinson's disease, spinal cord injury, severe diabetes, and severe hypertension etc;
5. Unable to complete motorized treadmill test at the speed of 2km/h;
6. Severe psychiatric disorder or cognitive impairment that prevent the understanding of the outcome evaluating questionnaires;
7. A history of lumbar surgery;
8. Have received acupuncture treatments in the previous 2 weeks;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who achieves at least 30% improvement in total walking distance from baseline. | Weeks 6 and 18
  The total walking distance is defined as the distance that participants forced to stop due to symptoms of neurogenic claudication or a time limit of 30 minutes during the motorized treadmill test (MTT).

SECONDARY OUTCOMES:
The proportion of participants who have at least 50% reduction from baseline in the average scores of buttocks and/or legs pain when walking, standing, or extending the back in the past week as measured by the Number Rating Scale (NRS). | Weeks 6,18 and 30
  Number Rating Scale (NRS) is a brief scale assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain. The minimum value is 0 points, and the maximum value is 10 points. The higher the score, the worse the result.
The proportion of participants who achieved at least 50% improvement in total walking distance from baseline. | Weeks 6 and 18
  The total walking distance is defined as the distance that participants forced to stop due to symptoms of neurogenic claudication or a time limit of 30 minutes during the MTT.
The change in total walking distance from baseline. | Weeks 6 and 18
  The total walking distance is defined as the distance that participants forced to stop due to symptoms of neurogenic claudication or a time limit of 30 minutes during the MTT.
The change in the time to first symptoms from baseline. | Weeks 6 and 18
  The time to first symptoms refers to the time when one or both legs experience pain, fatigue, abnormal sensations, and/or tightness during the MTT.
The change in the time to first moderate pain symptom from baseline. | Weeks 6 and 18
  The first moderate pain symptom refers to NRS score ≥4. Number Rating Scale (NRS) is a brief scale assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain. The minimum value is 0 points, and the maximum value is 10 points. The higher the score, the worse the result.
The change in final pain intensity from baseline. | Weeks 6 and 18
  When the subject reached their maximum distance, they were asked their NRS score, this was recorded as final pain intensity. Number Rating Scale (NRS) is a brief scale assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain. The minimum value is 0 points, and the maximum value is 10 points. The higher the score, the worse the result.
The change in recovery time from baseline. | Weeks 6 and 18
  Recovery time refers to time to return to baseline pain intensity after MTT.
The change in Modified Roland-Morris Disability Questionnaire (RMDQ) score from baseline. | Weeks 6,18 and 30
  Modified Roland-Morris Disability Questionnaire (RMDQ) is a reliable pain-specific functional status questionnaire which is easy and simple for patients to complete. The RMDQ includes 24 questions with a score range of 0-24. higher scores indicate more severe symptoms.
Changes from baseline in the average score of buttocks and/or legs pain when walking, standing, or extending the back as measured by the NRS in the previous 1 week. | Weeks 6,18 and 30
  Number Rating Scale (NRS) is a brief scale assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain. The minimum value is 0 points, and the maximum value is 10 points. The higher the score, the worse the result.
Changes in the average score of lower back pain when walking, standing, or extending the back as measured by the NRS in the previous 1 week from baseline. | Weeks 6,18 and 30
  Number Rating Scale (NRS) is a brief scale assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain. The minimum value is 0 points, and the maximum value is 10 points. The higher the score, the worse the result.
The change from baseline in the index score of European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L). | Weeks 6,18 and 30
  The European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L) includes five dimensions: Mobility, Self Care, Usual Activities, Pain or Discomfort, and Anxiety or Depression. Each dimension also includes five levels: no difficulty, slight difficulty, moderate difficulty, severe difficulty, and extreme difficulty. Each dimension has a high score of 5 and a low score of 1. The EQ-5D-5L index score can be calculated based on the choices made by the respondents on the five dimensions and five levels in the questionnaire.
The change from baseline in the domain scores (symptom severity and physical function) of Swiss Spinal Stenosis Questionnaire (SSSQ). | Weeks 6,18 and 30
  SSSQ include three domains, which are symptom severity, physical function and satisfaction with the treatment. Six questions in the symptom severity domain assess back, buttocks, legs or feet pain, pain frequency, numbness, weakness with scores ranging from 1 to 5 while one question assesses balance with scores ranging from 1, 3 and 5 and higher scores indicating worse symptoms. The physical function domain assesses walking distance and ability to walk for pleasure, shopping, and getting around the house or apartment and from the bathroom to the bedroom. This domain has five questions with scores ranging from 1 to 4, and higher scores indicate less satisfaction. For satisfactory domain, patients scoring 2.5 points or less are regarded as satisfied with the treatment.
The proportion of participants who are satisfied with the treatment based on the satisfaction domain of the SSSQ. | Weeks 6,18 and 30
  SSSQ include three domains, which are symptom severity, physical function and satisfaction with the treatment. Six questions in the symptom severity domain assess back, buttocks, legs or feet pain, pain frequency, numbness, weakness with scores ranging from 1 to 5 while one question assesses balance with scores ranging from 1, 3 and 5 and higher scores indicating worse symptoms. The physical function domain assesses walking distance and ability to walk for pleasure, shopping, and getting around the house or apartment and from the bathroom to the bedroom. This domain has five questions with scores ranging from 1 to 4, and higher scores indicate less satisfaction. For satisfactory domain, patients scoring 2.5 points or less are regarded as satisfied with the treatment.
The change from baseline in the total score of Hospital Anxiety and Depression Scale (HADS). | Weeks 6,18 and 30
  HADS is validated and standardized for measuring the state of anxiety and depression. HADS has 2 subscales with 14 items (7 items each), and a total score of 0 to 21 with 0 to 3 for each item.

OTHER OUTCOMES:
Expectance assessment | Baseline
  Expectancy of acupuncture will be recorded at baseline. Participants will be required to answer two questions: "In general, do you believe acupuncture is effective for treating the illness?" and "Do you think acupuncture will be helpful to improve your symptoms of LSS?"
Blinding assessment | Within 5 minutes after the either treatment in week 6
  Participants will be asked do you think you have received traditional acupuncture over the past 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China